CLINICAL TRIAL: NCT00562718
Title: A Pilot Safety And Feasibility Study Of Concurrent Capecitabine (Xeloda) And External Beam Irradiation In The Adjuvant Treatment Of High Risk Early Stage Breast Cancer.
Brief Title: Capecitabine and Radiation Therapy in Treating Patients With Nonmetastatic Breast Cancer After Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574761; SCCC-072004-004; ROCHE-SCCC-072004-004
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; male breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Capecitabine; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Surgery and Chemotherapy (Experimental): Eligible patients had undergone surgery and chemotherapy for high risk breast cancer, defined as either a T3 or T4 primary tumor, or N2 by either clinical or pathological criteria.
  Interventions: Drug: capecitabine; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: capecitabine
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x-rays to kill tumor cells. Capecitabine may also make tumor cells more sensitive to radiation therapy. Giving radiation together with capecitabine after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving capecitabine together with radiation therapy works in treating patients with nonmetastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety and feasibility of concurrent capecitabine and standard external-beam irradiation in patients with high-risk early stage breast cancer.

Secondary

* To determine the effects of concurrent treatment on cosmesis and wound healing at 1 year.
* To determine the short-term (1-year) risk of recurrence of breast cancer in these patients.

OUTLINE: This is a multicenter study.

Patients undergo external-beam radiotherapy once daily, 5 days a week and concurrently receive oral capecitabine twice daily, 5 days a week Monday through Friday, for approximately 6-7 weeks.

After completion of study therapy, patients are followed at approximately 1 week, 1 month, 6 months, and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive adenocarcinoma of the breast, meeting 1 of the following high-risk criteria:

  * T3 or T4 primary tumor
  * 4 or more involved axillary lymph nodes (N2 nodal stage)
* Completed surgical excision

  * No immediate reconstruction with autologous flap reconstruction

    * Patients having tissue expanders or implants placed prior to radiation may be enrolled at the physician's discretion
* No residual breast cancer

  * Microscopically positive margins are allowed if a re-excision is not felt to be clinically justified
* Candidate for radiotherapy

  * Must not require bilateral radiotherapy
* No metastatic (stage IV) breast cancer by AJCC staging criteria
* Hormone receptor status not specified
* No CNS disorders

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 6 months
* Karnofsky performance status 70-100%
* Menopausal status not specified
* Ambulatory
* Hemoglobin > 9 g/dL
* Platelet count > 100,000/mm³
* ANC > 1,500/mm³
* Serum AST, ALT, and alkaline phosphatase ≤ 2 times upper limit of normal (ULN)
* Total bilirubin normal
* Creatinine clearance > 50 mL/min
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception during study and for 30 days after the last study drug administration
* No serious, uncontrolled, concurrent infection(s)
* No diabetes with current or history of delayed wound healing or skin ulcers
* No autoimmune connective tissue disorder
* No prior unanticipated severe reaction to fluoropyrimidine therapy, known sensitivity to 5-fluorouracil, or known dihydropyrimidine dehydrogenase (DPD) deficiency
* No other carcinomas within the last five years except cured non-melanoma skin cancer and in-situ cervical cancer
* No clinically significant cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease, or cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months
* No other serious uncontrolled medical conditions that the investigator feels might compromise study participation, including any of the following:

  * Uncontrolled seizures
  * Psychiatric disability judged by the investigator to be clinically significant
* Physically intact upper gastrointestinal tract
* No malabsorption syndrome
* No uncompensated coagulopathy
* No patients whose breast size or body contour puts them at increased risk for skin desquamation from standard radiotherapy
* Able to read and speak English

PRIOR CONCURRENT THERAPY:

* Fully recovered from surgery and chemotherapy with completely healed surgical wounds
* At least 4 weeks since completion of prior chemotherapy regimen, excluding trastuzumab (Herceptin®)

  * Concurrent trastuzumab allowed at the physician's discretion
* More than 4 weeks since prior participation in any investigational drug study
* At least 4 weeks since prior and no concurrent sorivudine or brivudine
* More than 2 weeks since prior major surgery
* No prior capecitabine
* No prior radiotherapy to the chest or ipsilateral lymphatics
* No concurrent hormonal therapy during course of chemotherapy or radiation therapy
* No concurrent allopurinol or cimetidine
* Concurrent coumadin is allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only study
Enrollment: 50 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan P. Garwood, MD, Study Chair — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgery and Chemotherapy: Eligible patients had undergone surgery and chemotherapy for high risk breast cancer, defined as either a T3 or T4 primary tumor, or N2 by either clinical or pathological criteria.
  capecitabine
  adjuvant therapy
  radiation therapy
Period: Overall Study
Arm/Group | Surgery and Chemotherapy
Started | 50
Completed | 39
Not Completed | 11
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 2
Not completed — not stated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Surgery and Chemotherapy
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 52 [33 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 23
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39
masectomy [Count of Participants; unit: Participants] | 6
partial masectomy [Count of Participants; unit: Participants] | 22
neo-adjuvant [Count of Participants; unit: Participants] | 14
adjuvant [Count of Participants; unit: Participants] | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety
Description: Primarily Grade 1 and 2 toxicities attributable to capecitabine
Time Frame: 1 year
Population: Radiation given based on planned- 50.4cGy
Measure: Number; unit: percentage of participants
Arm/Group | Surgery and Chemotherapy
Number analyzed (Participants) | 28
percentage of participants | 12.6

2. Secondary Outcome: Cosmesis
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Surgery and Chemotherapy
Number analyzed (Participants) | 26
participants | 22

3. Secondary Outcome: Recurrence
Description: This population has aggressive disease with a high rate of recurrence and death within 1 year of completing radiation therapy
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Surgery and Chemotherapy
Number analyzed (Participants) | 28
percentage of participants | 14

ADVERSE EVENTS:
Arm/Group | Surgery and Chemotherapy
All-Cause Mortality (participants affected / at risk) | 6/39
Serious Adverse Events (participants affected / at risk) | 6/39
Other Adverse Events (participants affected / at risk) | 8/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery and Chemotherapy (N=39)
Radiation Dermatitis (Reproductive system and breast disorders) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery and Chemotherapy (N=39)
Diarrhea (Gastrointestinal disorders) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes